CLINICAL TRIAL: NCT03949192
Title: Efficacy of Hospital Traditional Chinese Medicine Preparation Kangliuwan for Recurrent Grade IV Glioma: A Prospective Exploratory Clinical Study
Brief Title: Efficacy of Kangliuwan for Recurrent Grade IV Glioma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Qingtang Lin, assistant director physician, Xuanwu Hospital, Beijing
Other Study IDs: LYS [2019] 027
Record Dates: First submitted 2019-05-11; First posted 2019-05-14 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Glioma of Brain; Recurrence
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Prospective Exploratory Clinical Study to explore the efficacy of Hospital Traditional Chinese Medicine Preparation Kangliuwan for Recurrent Grade IV Glioma.

ELIGIBILITY:
Inclusion Criteria:

1. The patient signed "informed consent" voluntarily;
2. The age of patient is between 18 and 80 years;
3. KPS score ≥40 ; The patient has normal liver and kidney function Normal heart function Better follow-up and compliance;

Exclusion Criteria:

1. The patient did not sign "informed consent" or signed unvoluntarily.
2. Non-glioma patients
3. Active infection
4. Human immunodeficiency virus (HIV) positive
5. Hepatitis C or hepatitis B infective
6. Pregnancy or breast-feeding women
7. Patients did not agree to use effective contraception during treatment and the following 3 months.
8. Patients also participated in other clinical studies.
9. The subjects researchers believe are not suitable for participation or completion of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recurrent grade IV glioma patients and conventional treatment is invalid.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-06-28 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes in tumor volume | 3 months
  the volume of tumor decreased after taking Kangliuwan

CONTACTS AND LOCATIONS:
Overall Officials: Qingtang Lin, M.D., Ph.D., Study Chair — Xuanwu Hospital, Beijing; Xiaolan Lin, M.D., Principal Investigator — Xuanwu Hospital, Beijing; Ling Chen, M.D., Principal Investigator — The General Hospital of People's Liberation Army (301 hospital)
Locations (1):
- Xuanwu Hospital, Beijing, Beijing Municipality, China